CLINICAL TRIAL: NCT01615263
Title: Isolated Lung Collapse in Two Stages With Bronchial Blocker: Comparison With Double Lumen Tube
Brief Title: Lung Collapse With Bronchial Blocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Full clinical professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IUCPQ 20784
Record Dates: First submitted 2012-05-25; First posted 2012-06-08 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Video-assisted Thoracoscopic Surgery; Lung Isolation Device; One-lung Ventilation; Double Lumen Endotracheal Tube; Bronchial Blocker
Keywords: Video-assisted thoracoscopic surgery (VATS); One lung ventilation; Bronchial blocker; Lung collapse; Double lumen tube
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double lumen tube (Active Comparator): Lung isolation with a left double lumen tube (BronchoCath, Mallinckrodt Medical, Cornamaddy, Athlone, Westmeath, Ireland.
  Interventions: Device: Lung isolation device
- Bronchial blocker (Active Comparator): Lung isolation with a bronchial blocker with the inner channel closed (Fuji Uniblocker 9F, Fuji System Corporation, Tokyo, 113-0033, Japan) inserted via a 8.0 mm simple lumen endotracheal tube.
  Interventions: Device: Lung isolation device

INTERVENTIONS:
Device: Lung isolation device — Lung isolation for one-lung ventilation with a left double lumen tube
  Other Names: BronchoCath, Mallinckrodt Medical
  Arms: Double lumen tube
Device: Lung isolation device — Lung isolation for one-lung ventilation with a bronchial blocker inserted through a 8.0 mm simple lumen endotracheal tube
  Other Names: Fuji Uniblocker 9 French
  Arms: Bronchial blocker

SUMMARY:
Lung isolation is frequently used during thoracic surgery. Two techniques are principally used: the double lumen tube (DLT) and the bronchial blocker (BB). BB is easy to use but its reputation is darken by the need of multiple repositioning during surgery and especially by a slower lung collapse than the DLT. Reading recent literature on the subject and according to the vast experience of numerous hospital centers, it seems that the slowness of lung collapse remains without any solution. This slowness in lung deflation is detrimental to the initiation of video-assisted thoracoscopy surgery (VATS) and could be exacerbated in chronic obstructive disease (COPD) patients. For this reason, BB use is discredited in numerous centers. However, at IUCPQ, the investigators rarely observe slow lung collapse when BB are used. For many years, the investigators have used a systematic denitrogenation of the lung before the initiation of one lung ventilation (OLV). Furthermore, when the patient is positioned in lateral decubitus, the investigators impose an apnea period of about 30 seconds to favor collapse of the isolated lung before inflating the cuff. This apnea is always limited by the occurrence of oxygen desaturation (≤97%). The investigators also proceed to a second period of apnea of 30 seconds associated to a deflated BB's cuff at the pleural opening. Subsequently, the investigators inflate the BB's cuff to obtain definitive lung isolation. The investigators hypothesis is that the use of two apnea periods, when isolating the lung with a BB, will allow the same quality of surgical exposure at 0, 5, 10 and 20 minutes post opening of the pleura, compared to the one obtained with a DLT. The main objective of this study is first to compare the delay between the initiation of OLV and complete lung collapse obtained with BB and DLT, in two groups of patients undergoing VATS. Secondary objectives are: 1) to evaluate the quality of surgical exposure associated to the level of lung collapse, 2) to evaluate the quality of surgical exposure through the video camera, 3) to collect surgeons' opinion regarding the device (BB or DLT) that they thought was used during surgery. After obtaining institutional review board (IRB) approval, the investigators propose a study of 40 patients undergoing an elective VATS at the Institut universitaire de cardiologie et pneumologie de Québec (IUCPQ) involving an one lung ventilation. They will have to be 18 years old or more, to read, understand and sign an informed consent at their pre-operative evaluation. This study will be prospective, randomized, and blind to thoracic surgeons.

DETAILED DESCRIPTION:
Background:

Lung isolation is frequently used during thoracic surgery. Two techniques are principally used: the double lumen tube (DLT) and the bronchial blocker (BB). Today, the thoracic surgical technique with more perspective is the video-assisted thoracoscopy surgery (VATS), which requires an effective lung isolation technique

The DLT is the one that is widely used by the vast majority of anesthesiologists. It has been introduced in the eighties in its actual version of polyvinyl chloride. Its positioning with a fibrobronchoscope (FOB) is well established. Its efficiency is reproducible and it is used without major complication. Its use is limited in the presence of difficult airway.

The BB had appeared in its modern form at the end of the 1990. It is easy to use but its reputation is darken by the need of multiple repositioning during surgery and especially by a slower lung collapse than the DLT. The collapse of the isolated lung is the result of denitrogenation atelectasis and the draining of isolated lung through the inner channel of the BB. The diameter and the length of the internal channel vary depending of the model. The BB inner channel is very much smaller (Cook's Arndt: 1.3 mm; Cook's Cohen: 1.6 mm and Fuji's Uniblocker: 2.0 mm) than the lumen of a DLT, which varies from 6 to 9 mm (for a 35 to a 41 Fr tube).

A comparative study published in 2003 by Campos demonstrated results in favor of the inner channel draining hypothesis. Authors showed that the lung collapse with the Arndt BB is longer than with the Uniblocker BB or the BronchoCath DLT and that it needs more suction through the inner channel (p>0.06). The limitation of this report is that the number of thoracotomies and of video-assisted thoracoscopies surgery (VATS) was not mentioned. Furthermore, the side of surgery was not specified. This point is very important since the inflated cuff of a BB located into the right main bronchus may obstruct the origin the right upper lobe, and consequently impair its collapse.

In 2009, with a series of 45 thoracotomies and 22 VATS, Narayanaswamy and Slinger demonstrated that when both lung isolation and one lung ventilation (OLV) are started early, meaning immediately post-induction and intubation in dorsal decubitus position, and continuously maintained until the pleural is opened. Similar surgical exposure at 10 and 20 minutes post pleural opening was obtained with all three modern BB as with left DLT. In this report, the duration of the lung isolation period and of the one lung ventilation was not specified. We presume that this length was over 20 or 30 minutes before pleural opening, which created a lung collapse by denitrogenation, as shown by a later publication by the same research team. An early -20 cmH2O suction (at the start of OLV) through either a DLT or a Cohen's BB improved lung collapse quality compared to a late application (20 min after pleural opening). This advantage was not demonstrated with the Arndt BB or the Fuji's. Another limitation of this study is that it was done with only left unilateral surgeries to avoid inflating the BB cuff into the right main bronchus. This choice creates an important selection bias since these results cannot be applied to a universal use of BB.

In 2009, Ko and Slinger also published the following: the use of a fraction of inspired oxygen (FiO2) of 1.0 (denitrogenation) while ventilating before the initiation of OLV through a DLT gives a better surgical exposure at 10 and 20 minutes compared to a FiO2 of 0.4. These results are from 4 VATS and 100 thoracotomies.

Early initiation of OLV in dorsal decubitus is not recommended by any author for the following reasons: an additional OLV period of 15 to 30 minutes is not beneficial for the patient if desaturation occurs. Moreover, mobilization of patient in lateral decubitus could lead to complications related to an inflated BB. In fact, proximal movement of the BB's cuff can completely obstruct the trachea. There is also a risk of trauma to the airway. Note that these risks are theoretical since they were note described in this context. Since it is recommended to proceed to lung isolation when the patient in positioned in lateral decubitus, it is not surprising that these complications are not reported in the literature.

Reading recent literature on the subject and according to the vast experience of numerous hospital centers, it seems that the slowness of lung collapse remains without any solution. This slowness in lung deflation is detrimental to the initiation of VATS and could be exacerbated in COPD patients. For this reason, BB use is discredited in numerous centers.

However, at IUCPQ, the investigators rarely observe slow lung collapse when BB are used. For many years, the investigators have used a systematic denitrogenation of the lung before the initiation of OLV. Furthermore, when the patient is positioned in lateral decubitus, the investigators impose an apnea period of about 30 seconds to favor collapse of the isolated lung before inflating the cuff. This apnea is always limited by the occurrence of O2 desaturation (≤97%). The investigators also proceed to a second period of apnea of 30 seconds associated to a deflated BB's cuff at the pleural opening. Subsequently, the investigators inflate the BB's cuff to obtain definitive lung isolation.

Actual literature does not allow the anesthesiologists to conclude clearly on a choice of bronchial blocker. Thus, the investigators propose a study that will add up to essential data to make a better choice of lung isolation device.

Hypothesis:

The investigators hypothesis is that the use of two apnea periods, when isolating the lung with a BB, will allow the same quality of surgical exposure at 0, 5, 10, and 20 minutes post opening of the pleura compared to the one obtained with DLT. The investigators will use Fuji's BB and occlude its internal channel to be able to extrapolate the investigators results with other BB that are actually on the market.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* elective video-assisted thoracoscopy
* one lung ventilation

Exclusion Criteria:

* Difficult mask ventilation
* planned difficult intubation
* use of a right double lumen tube
* severe COPD (VEMS < 50% and Tiffeneau < 50% of the predicted values)
* asthma (instable <1 year)
* bulla disease
* pleural disease
* previous ipsilateral thoracic surgery
* thoracic radiotherapy
* significant systemic co-morbidity
* active or chronic pulmonary infection
* fibrosis, other interstitial diseases
* endobronchial mass
* right upper lobe bronchus at the pericarinal level (preoperative or at the first FOB under anesthesia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Campos JH, Kernstine KH. A comparison of a left-sided Broncho-Cath with the torque control blocker univent and the wire-guided blocker. Anesth Analg. 2003 Jan;96(1):283-9, table of contents. doi: 10.1097/00000539-200301000-00056. PMID 12505967
- [Background] Ko R, McRae K, Darling G, Waddell TK, McGlade D, Cheung K, Katz J, Slinger P. The use of air in the inspired gas mixture during two-lung ventilation delays lung collapse during one-lung ventilation. Anesth Analg. 2009 Apr;108(4):1092-6. doi: 10.1213/ane.0b013e318195415f. PMID 19299766
- [Background] Narayanaswamy M, McRae K, Slinger P, Dugas G, Kanellakos GW, Roscoe A, Lacroix M. Choosing a lung isolation device for thoracic surgery: a randomized trial of three bronchial blockers versus double-lumen tubes. Anesth Analg. 2009 Apr;108(4):1097-101. doi: 10.1213/ane.0b013e3181999339. PMID 19299767
- [Background] Brodsky JB. Lung separation and the difficult airway. Br J Anaesth. 2009 Dec;103 Suppl 1:i66-75. doi: 10.1093/bja/aep262. PMID 20007992
- [Background] Fortier G, Cote D, Bergeron C, Bussieres JS. New landmarks improve the positioning of the left Broncho-Cath double-lumen tube-comparison with the classic technique. Can J Anaesth. 2001 Sep;48(8):790-4. doi: 10.1007/BF03016696. PMID 11546721
- [Derived] Bussieres JS, Somma J, Del Castillo JL, Lemieux J, Conti M, Ugalde PA, Gagne N, Lacasse Y. Bronchial blocker versus left double-lumen endotracheal tube in video-assisted thoracoscopic surgery: a randomized-controlled trial examining time and quality of lung deflation. Can J Anaesth. 2016 Jul;63(7):818-27. doi: 10.1007/s12630-016-0657-3. Epub 2016 May 2. PMID 27138896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April to October 1st 2012, 111 patients were assessed for inclusion criteria. 71 patients were not included and 40 were enrolled at their pre-operative visit to the thoracic surgery department.
Pre-assignment Details: No enrolled patient was excluded from the study prior to the randomization.
Groups:
- Double Lumen Tube: Lung isolation with a left double lumen tube (BronchoCath, Mallinckrodt Medical, Ireland.)
- Bronchial Blocker: Lung isolation with a bronchial blocker with the inner channel closed (Fuji Uniblocker 9 Fr, Fuji System Corporation, Tokyo, 113-0033, Japan) inserted via a 8.0 mm simple lumen endotracheal tube.
Period: Overall Study
Arm/Group | Double Lumen Tube | Bronchial Blocker
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Post-randomization exclusion | 0 | 2

BASELINE CHARACTERISTICS:
Population: Comparability test was calculated with a difference of 15% to allow a mean collapse time of 18 min with an alpha of 0.05 and power of 0.90. Sample size was estimated at 18 patients. 20 patients per group were randomized. 2 patients were excluded: 1 for tracheal origin of right upper lobe (RUL) bronchus, 1 for severe desaturation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Lumen Tube | Bronchial Blocker | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (18.2) | 61.9 (7.5) | 62.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Time to Obtain Complete Lung Collapse
Description: For patients intubated with double lumen tube (DLT), clamping of the ipsilateral lumen without continuous positive airway pressure (CPAP) on the isolated lung will be done to allow lung collapse. The timer will be started at this moment and stopped 20 minutes after pleural opening. For patients of the bronchial blocker (BB) group, the first apnea period will of 30 seconds, keeping a pulse oximetry (SpO2) always over 97%, and under direct visualization with the FOB. Afterward, the cuff will be reflated and the timer will be started at this moment and stopped 20 minutes after pleural opening. For both groups, time of total lung collapse will be measured.
Time Frame: From the beginning of one lung ventilation to 20 minutes after pleural opening
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Double Lumen Tube: Lung isolation with a left double lumen tube (BronchoCath, Mallinckrodt Medical, Cornamaddy, Athlone, Westmeath, Ireland.)
Arm/Group | Double Lumen Tube | Bronchial Blocker
Number analyzed (Participants) | 20 | 18
minutes | 47.8 (35.9) | 32.5 (11.8)

2. Secondary Outcome: Quality of Lung Collapse
Description: Assessment of lung collapse by the thoracic surgeon at 0, 5, 10 and 20 minutes after pleural opening.Visual analog scale of the quality of lung collapse will be assessed as the following:
  1. No lung collapse
  2. Partial lung collapse, not satisfactory
  3. Partial lung collapse, satisfactory
  4. Complete lung collapse
Time Frame: From pleural opening to 20 minutes after
Measure: Number; unit: percentage of patients
Arm/Group | Double Lumen Tube | Bronchial Blocker
Number analyzed (Participants) | 20 | 18
percentage of patients
  Time 0, No lung collapse | 10 | 6
  Time 0, Partial lung collapse, not satisfactory | 45 | 17
  Time 0, Partial lung collapse, satisfactory | 30 | 55
  Time 0, Complete lung collapse | 15 | 22
  Time 5 min, No lung collapse | 5 | 0
  Time 5 min, Partial lung collapse not satisfactory | 10 | 6
  Time 5 min Partial lung collapse, satisfactory | 65 | 39
  Time 5 min Complete lung collapse | 20 | 55
  Time 10 min, No lung collapse | 0 | 0
  Time 10 min Partial lung collapse not satisfactory | 10 | 0
  Time 10 min Partial lung collapse, satisfactory | 60 | 33
  Time 10 min Complete lung collapse | 30 | 67
  Time 20 min, No lung collapse | 0 | 0
  Time 20 min Partial lung collapse not satisfactory | 5 | 0
  Time 20 min Partial lung collapse, satisfactory | 50 | 22
  Time 20 min Complete lung collapse | 45 | 78

3. Secondary Outcome: Opinion on the Device
Description: 20 minutes after pleural opening, the thoracic surgeon will give his opinion on the lung isolation device that was used on his patient (double lumen tube or bronchial blocker).
Time Frame: 20 minutes after pleural opening
Measure: Number; unit: percentage of right guess/opinion
Arm/Group | Double Lumen Tube | Bronchial Blocker
Number analyzed (Participants) | 20 | 18
percentage of right guess/opinion | 50 | 22.2

4. Secondary Outcome: Use of Suction to Facilitate Lung Collapse
Time Frame: Up to 5 minutes after surgery
Measure: Number; unit: participants
Arm/Group | Double Lumen Tube | Bronchial Blocker
Number analyzed (Participants) | 20 | 18
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Double Lumen Tube | Bronchial Blocker
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes